CLINICAL TRIAL: NCT01968369
Title: Effects of Tomato Sauce on Endothelial Dysfunction Induced by a High Fat Meal in Healthy Subjects
Acronym: VRPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Cristiano Fava, MD, PhD, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: VRPM_Tomato_and_endothelium
Record Dates: First submitted 2013-10-16; First posted 2013-10-24 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Endothelial Dysfunction
Keywords: flow mediated vasodilatation; tomato; arterial stiffness; lycopene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tomato sauce (+/- high fat meal) (Active Comparator): 80 gr for 7 days= total load 560 mg (+/- high fat meal)
  Interventions: Dietary Supplement: tomato sauce
- diet without tomato (+/- high fat meal) (Placebo Comparator): diet without tomato (+/- high fat meal)
  Interventions: Dietary Supplement: tomato sauce

INTERVENTIONS:
Dietary Supplement: tomato sauce — We are randomising healthy men (N=14-28) to consume a high fat meal either with or without tomato sauce (80 gr) in a cross-over design with a 7 days wash-out period. During the week before the study, all the subjects will be maintained in a low fibers diet and only subjects randomized to tomatoes will receive a daily dose of 80 mg of tomato sauce (80 gr for 7 days= total load 560 mg).

SUMMARY:
Several epidemiological and intervention studies suggest that a high dietary intake of tomatoes is associated with lower risk of cardiovascular disease (CVD), while, low intake is associated with an increased incidence of CVD. This beneficial effects have been attributed especially to lycopene, an antioxidant present in high concentration within tomatoes but other substances could be of importance.

Endothelial dysfunction is an early marker of atherosclerosis leading to CVD. The aim of the present study is therefore to investigate whether consumption of tomato products ameliorates peripheral endothelial function, triggered by a high fat meal, in human volunteers in a randomised, crossover dietary intervention study.

Study design:

Investigators are randomising healthy men (N=14-28) to consume a high fat meal either with or without tomato sauce (80 gr) in a cross-over design with a 7 days wash-out period. During the week before the study all the subjects will be maintained in a low fibers diet and only subjects randomized to tomatoes will receive a daily dose of 80 mg of tomato sauce (80 gr for 7 days= total load 560 mg).

We hypothesize that tomato sauce can improve the deleterious effects of a high fat meal on vascular function.

DETAILED DESCRIPTION:
Several epidemiological and intervention studies suggest that a high dietary intake of tomatoes is associated with lower risk of cardiovascular disease (CVD), while, low intake is associated with an increased incidence of CVD. This beneficial effects have been attributed especially to lycopene, an antioxidant present in high concentration within tomatoes but other substances could be of importance.

Endothelial dysfunction is an early marker of atherosclerosis leading to CVD. The aim of the present study is therefore to investigate whether consumption of tomato products ameliorates peripheral endothelial function, triggered by a high fat meal, in human volunteers in a randomised, crossover dietary intervention study.

Study design:

Investigators are randomising healthy men (N=14-28) to consume a high fat meal either with or without tomato sauce (80 gr) in a cross-over design with a 7 days wash-out period. During the week before the study all the subjects will be maintained in a low fibers diet and only subjects randomized to tomatoes will receive a daily dose of 80 mg of tomato sauce (80 gr for 7 days= total load 560 mg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men,
* without overt risk factors for CVD (see exclusion criteria);
* age range 28 ±10 years;
* BMI between 19-27 Kg/m2

Exclusion Criteria:

* Previous cardiovascular events, kidney failure (serum creatinine ≥1,5 mg/dl), arterial blood pressure ≥140/90mmHg or diagnosed hypertension; chronic inflammatory or neoplastic diseases, diabetes mellitus or impaired fasting glucose (glucose ≥110 mg/dL), hypercholesterolemia (total cholesterol ≥240 mg/dl or anti-lipemic medication use), current smoking, antihypertensive medications; use of antioxidant drugs or NSAIDs or COXIBs; food allergy to tomato or other components of the high fat diet.

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilatation (FMD) | change in FMD 2 and 3.5 hour after a high fat meal
  Endothelial function as measured non-invasively by ultrasound (LogiQ P5 pro, GE Healthcare) using the "Flow Mediated Dilatation" (FMD) technique with the aid of a dedicated hardware (Multimedia Video Engine II (MVE2) DSP Lab., Pisa CNR, Italy).

SECONDARY OUTCOMES:
Arterial stiffness measured as Stiffness Index (SI), Carotid distensibility (CD) | change in SI and CD 2 and 3.5 hour after a high fat meal
  systemic and local arterial stiffness measured by digital photoplethysmography (PulseTracePT1000 - MicroMedical Ltd) and by carotid ultrasound (LogiQ P5 pro, GE Healthcare) with the aid of a dedicated hardware (Multimedia Video Engine II (MVE2) DSP Lab., Pisa CNR, Italy).
inflammatory cytokines | chnage in inflammatory cytokines 2 and 3.5 hour after a high fat meal
blood pressure | change in blood pressure 2 and 3.5 hour after a high fat mealeal
  office blood pressure measured by a semiautomatic oscillometric device (TM-2501, A&D instruments Ltd)

OTHER OUTCOMES:
plasma level of lycopene and other substances contained in tomatoes. | change 2 and 3.5 hour after a high fat meal
glucose and lipid | change 2 and 3.5 hour after a high fat meal
  glucose and lipid variation

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Fava, M.D.; PhD, Principal Investigator — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy